CLINICAL TRIAL: NCT03625284
Title: Oral Dietary Fucoxanthin Rich Supplement for Liver Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Algatechnologies Ltd. (Industry)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Clinical protocol FUCO 02
Record Dates: First submitted 2018-07-02; First posted 2018-08-10 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Non Alcoholic Fatty Liver
Keywords: fucoxanthin; microalgae; non alcoholic fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — fucoxanthin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fucovital (Experimental): capsules of a dietary supplement rich with fucoxanthin from microalgae extract
  Interventions: Dietary Supplement: FucoVital
- Placebo (Placebo Comparator): capsules of an edible oil
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: FucoVital

INTERVENTIONS:
Dietary Supplement: Placebo — Edible oil
  Arms: Placebo
Dietary Supplement: FucoVital — Microalgae oil extract
  Other Names: fucoxanthin

SUMMARY:
Blind, placebo-controlled study testing the hypothesis that oral dietary supplement rich with fucoxanthin will decrease biochemical clinical markers related to liver health.

DETAILED DESCRIPTION:
Six month supplementation

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults > 18 years
* Willing to sign an informed consent to participate in the study.
* Non-smokers.
* Blood results above the normal range in hepatic function testing consisting of panels containing ALT, AST, ALP, total bilirubin and albumin and abdominal ultrasonography.
* Over-weight (BMI ≥ 27 kg/m2) who fulfill the criteria of the National Cholesterol Education Program (NCEP) metabolic syndrome.

Exclusion Criteria:

* Pregnancy.
* Presence of gastrointestinal or mental disorders, diabetes mellitus, alcohol abuse, weight-loss treatment, bariatric surgery, unusual diets (vegetarian, vegan), daily usage of antioxidants dietary supplements at the last 4 months (for subjects in stage 2 of the study).
* Serious medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-10 (Estimated); Primary Completion 2019-09-10 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
Liver function test: Serum Alanine transaminase (ALT) | week 0,12,24
  Change from baseline of liver enzymes
Liver function test: Aspartate transaminase (AST) | week 0,12,24
  Change from baseline of liver enzymes

SECONDARY OUTCOMES:
Liver function test:Blood gamma-glutamyl transferase (GGT) | week 0,12,24
  change from baseline
Liver function test:Blood albumin | week 0,12,24
  change from baseline
Liver function test: Blood bilirubin | week 0,12,24
  change from baseline
Hepatic steatosis | 0, 24 week
  Change from baseline by ultrasound
Weight | week 0,12,24
  Change from baseline
Waist circumference | week 0,12,24
  Change from baseline
Serum lipid profile | week 0,12,24
  Change from baseline total cholesterol, triglycerides, low density lipoprotein (LDL) (HDL) fractions
Blood glucose status | week 0,12,24
  Change from baseline of HbA1c
Inflammation | week 0,12,24
  Change from baseline of CRP
Kidney function test: serum creatinine | week 0,12,24
  Change from baseline
Kidney function test: Glomerular Filtration Rate(GFR) | week 0,12,24
  Change from baseline
Kidney function test: Blood Urea Nitrogen | week 0,12,24
  Change from baseline
Dietary supplement level in the blood | week 0,6 or 12,24
  Determination of Fucoxanthin metabolite in plasma by LC-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Haim Shirin, Prof., Principal Investigator — Director Institute of Gastroenterolgy, Liver Diseases and Nutrition

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang M, Xuan Z, Wang Q, Yan S, Zhou D, Naman CB, Zhang J, He S, Yan X, Cui W. Fucoxanthin has potential for therapeutic efficacy in neurodegenerative disorders by acting on multiple targets. Nutr Neurosci. 2022 Oct;25(10):2167-2180. doi: 10.1080/1028415X.2021.1926140. Epub 2021 May 15. PMID 33993853